CLINICAL TRIAL: NCT00343798
Title: A Pilot Study to Evaluate the Co-infusion of Ex Vivo Expanded Umbilical Cord Blood Progenitors With an Unmanipulated Cord Blood Graft in Patients Undergoing Umbilical Cord Blood Transplantation for Hematologic Malignancies
Brief Title: A Pilot Study to Evaluate the Co-Infusion of Ex Vivo Expanded Cord Blood Cells With an Unmanipulated Cord Blood Unit in Patients Undergoing Cord Blood Transplant for Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2044.00; NCI-2010-00236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R43HL106868 (NIH); R24HL074445 (NIH); RC2HL101844 (NIH)
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Previously Treated Myelodysplastic Syndromes; Prolymphocytic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Childhood Lymphoblastic Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage II Childhood Lymphoblastic Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Childhood Lymphoblastic Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Leukemia, Prolymphocytic; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine phosphate; Cyclosporine; Mycophenolic Acid; Biopsy; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (umbilical cord blood transplant) (Experimental): MYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -8 to -6 and cyclophosphamide IV on days -7 and -6. Patients undergo TBI BID on days -4 to -1.
  TRANSPLANTATION : Patients undergo double-unit umbilical cord blood transplantation comprising unmanipulated umbilical cord blood unit IV over 20-30 minutes, and 4-6 hours later patients receive ex vivo-expanded umbilical cord blood cells IV over 30 minutes on day 0.
  GRAFT-VERSUS-HOST-DISEASE PROPHYLAXIS: Patients receive cyclosporine IV every 8 or 12 hours on days -3 to 100, followed by a taper to at least day 180. Patients also receive MMF IV every 8 hours on days -3 to 5 and then PO, if tolerated, on days 6-30.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: ex-vivo umbilical cord blood expansion; Procedure: double-unit umbilical cord blood transplantation; Procedure: biopsy; Other: immunologic technique; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclosporine — Given IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Other: ex-vivo umbilical cord blood expansion — Undergo double-unit umbilical cord blood transplantation
Procedure: double-unit umbilical cord blood transplantation — Undergo double-unit umbilical cord blood transplantation
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Other: diagnostic laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I multicenter feasibility trial is studying the safety and potential efficacy of infusing ex vivo expanded cord blood progenitors with one unmanipulated umbilical cord blood unit for transplantation following conditioning with fludarabine, cyclophosphamide and total body irradiation (TBI), and immunosuppression with cyclosporine and mycophenolate mofetil (MMF) for patients with hematologic malignancies. Chemotherapy, such as fludarabine and cyclophosphamide, and TBI given before an umbilical cord blood transplant stops the growth of leukemia cells and works to prevent the patient's immune system from rejecting the donor's stem cells. The healthy stem cells from the donor's umbilical cord blood help the patient's bone marrow make new red blood cells, white blood cells, and platelets. It may take several weeks for these new blood cells to grow. During that period of time, patients are at increased risk for bleeding and infection. Faster recovery of white blood cells may decrease the number and severity of infections. Studies have shown that counts are more likely to recover more quickly if increased numbers of cord blood cells are given with the transplant. We have developed a way of growing or "expanding" the number of cord blood cells in the lab so that there are more cells available for transplant. We are doing this study to find out whether or not giving these expanded cells along with one unexpanded cord blood unit is safe and if use of expanded cells can decrease the time it takes for white blood cells to recover after transplant. We will study the time it takes for blood counts to recover, which of the two cord blood units makes up the patient's new blood system, and how quickly immune system cells return

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the safety and toxicity when ex vivo expanded cord blood cells are co-infused with a second non-human leukocyte antigen (HLA)-identical cord blood graft following myeloablative therapy in patients with hematologic malignancies.

II. Examine the in vivo persistence of the ex vivo expanded cord blood cells. The kinetics and durability of hematopoietic reconstitution (time to engraftment defined as the first of 2 consecutive days in which the absolute neutrophil count [ANC] > 500) will be determined and the relative contribution to engraftment of the expanded cord blood cells and the unmanipulated cord blood cells in early and long-term engraftment will be determined by donor chimerisms.

SECONDARY OBJECTIVES:

I. Estimate the incidence and severity of acute and chronic graft-versus-host disease (GVHD) in patients receiving Notch-expanded cord blood cells.

II. Estimate the incidence of transplant related mortality at day 100.

III. Estimate the incidence of malignant relapse and probabilities of overall and event-free survival at 1 and 2 years post transplant.

IV. Obtain preliminary data on the phenotype and function of immune cells recovering in patients receiving expanded and unmanipulated cord blood grafts.

V. Obtain feasibility data on overnight shipment of ex vivo expanded progenitor cells for infusion in patients are distant sites.

OUTLINE:

MYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine intravenously (IV) over 1 hour on days -8 to -6 and cyclophosphamide IV on days -7 and -6. Patients undergo TBI twice daily (BID) on days -4 to -1.

TRANSPLANTATION : On Day 0, patients undergo double-unit umbilical cord blood transplantation which includes the infusion of one unmanipulated (not expanded) cord blood unit followed 4 hours later by infusion of one ex vivo-expanded cord blood unit.

GRAFT-VERSUS-HOST-DISEASE PROPHYLAXIS: Patients initially receive cyclosporine IV beginning on day -3. Cyclosporine may be given orally when the patient can tolerate oral medications and has a normal gastrointestinal transit time. Cyclosporine is given until day 100, and may taper on day 101 if there is no graft versus host disease. Patients also receive MMF IV on days -3 to 5 and then may receive oral MMF beginning day 6 to 30. MMF is stopped at Day 30 or 7 days after engraftment, whichever day is later, if no acute GVHD.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has no existing 0-1 HLA-A, B, C, DRB1 and DQB1 matched related donor
* Acute Myeloid Leukemia:

  * High risk first complete remission (CR1) as evidenced by preceding myelodysplastic syndromes (MDS), high risk cytogenetics (for example, monosomy 5 or 7, or HR as defined by referring institution treatment protocol), >= 2 cycles to obtain complete remission (CR), erythroblastic or megakaryocytic leukemia; >= second complete remission (CR2);
  * All patients must be in CR as defined by hematologic recovery and < 5% blasts by morphology within the bone marrow and a cellularity of >= 15%;
  * Patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry (< 5% blasts) and, recovery of peripheral blood counts with no circulating blasts, may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures
* Acute lymphoblastic leukemia:

  * High risk CR1 (for example, but not limited to: t(9;22), t(1;19), t(4;11) or other mixed-lineage leukemia (MLL) rearrangements, hypodiploid);
  * > 1 cycle to obtain CR;
  * >= CR2;
  * All patients must be in CR as defined by hematologic recovery and < 5% blasts by morphology within the bone marrow and a cellularity of >= 15%;
  * Patients in which adequate marrow/biopsy specimens can not be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry (< 5% blasts) and, recovery of peripheral blood counts with no circulating blasts, may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures
* Chronic Myelogenous Leukemia:

  * Patients in blast crisis (BC) must receive therapy and must achieve accelerated phase (AP)/chronic phase (CP) in order to be eligible (patients who remain in BC are not eligible);
  * If in first chronic phase, patient must have failed or be intolerant to imatinib mesylate
* Myelodysplasia (MDS):

  * International Prognostic Scoring System (IPSS) Int-2 or high risk (Refractory anemia with excess blasts [RAEB], refractory anemia with excess blasts in transformation [RAEBt]) or refractory anemia with severe pancytopenia or high risk cytogenetics;
  * Blasts must be < 10% morphologically in representative bone marrow aspirate (obtained < 2 weeks from enrollment)
* Lymphoblastic lymphoma, Burkitt's lymphoma, and other high-grade non-Hodgkin lymphoma (NHL) after initial therapy if stage III/IV in first partial remission (PR1) or after progression if stage I/II < 1 year; Stage III/IV patients are eligible after progression in complete response (CR)/partial response (PR)
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, lymphoplasmacytic lymphoma or follicular lymphoma that have progressed after at least two different prior therapies; patients with bulky disease (nodal mass greater than 5 cm) should be considered for debulking chemotherapy before transplant (these patients must be presented at Patient Care Conference [PCC] prior to enrollment given potential competing eligibility on autotransplant protocols)
* Mantle-cell lymphoma, prolymphocytic leukemia: Eligible after initial therapy in >= CR1 or >= PR1
* Large cell NHL > CR2/ > PR2:

  * Patients in CR2/PR2 with initial short remission (< 6 months) are eligible;
  * These patients must be presented at PCC prior to enrollment given potential competing eligibility on autotransplant protocols
* Multiple myeloma beyond PR2: Patients with chromosome 13 abnormalities, first response lasting less than 6 months, or beta-2 microglobulin > 3 mg/L, may be considered for this protocol after initial therapy
* Serum creatinine =< 2.0 mg/dL (adults) and creatinine clearance > 60 ml/min (pediatrics)
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, histology, and the degree of portal hypertension; patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL and symptomatic biliary disease will be excluded
* Diffusing capacity of the lung for carbon monoxide corrected (DLCOcorr) > 50% normal
* Left ventricular ejection fraction >= 45% or shortening fraction > 26%
* Karnofsky score >= 70% (adults) or Lansky score >= 50% (pediatrics)

Exclusion Criteria:

* Acute leukemia in relapse (>= 5% marrow blasts by morphology)
* Active central nervous system (CNS) leukemia involvement at the time of study enrollment (cerebrospinal fluid with > 5 white blood cells (WBC)/mm^3 AND malignant cells on cytospin)
* Chemotherapy refractory large cell lymphoma and high grade NHL (progressive disease after > 2 salvage regimens)
* Female patients who are pregnant or breastfeeding
* Karnofsky performance status < 70% (adults) or Lanksy score < 50% (pediatrics)
* Prior autologous or allogeneic stem cell transplant with myeloablative preparative regimen (If =< 18 years old, prior myeloablative transplant within the last 6 months)
* Uncontrolled viral, or bacterial infection at the time of study enrollment
* Active or recent (prior 6 months) invasive fungal infection without ID consult and approval
* Seropositive for human immunodeficiency virus (HIV)
* Consenting 5 of 6 or 6 of 6 HLA-matched related donor available
* Unable to provide informed consent
* Use of any other experimental drug within 28 days of baseline

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2006-04; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Severe (grades 3 and 4) acute GVHD | Up to day 100
Grade greater than or equal to 3 infusional toxicity | Day 0
Graft failure as defined by failure to achieve ANC greater than or equal to 500/mm^3 of donor origin | By day +42

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Delaney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington